CLINICAL TRIAL: NCT01951300
Title: 68Ga-Citrate Positron Emission Tomography (PET) of Healthy Volunteers
Brief Title: 68Ga-Citrate PET of Healthy Volunteers
Acronym: SITRAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Anne Roivainen, professor, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 167/2013
Record Dates: First submitted 2013-09-03; First posted 2013-09-26 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
MeSH Terms: interventions — gallium citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gallium-68 citrate (Other): Intravenous bolus injection of 200 MBq of Gallium-68 citrate
  Interventions: Other: Gallium-68 citrate

INTERVENTIONS:
Other: Gallium-68 citrate — Single intravenous bolus injection of 200 MBq of Gallium-68 citrate radiopharmaceutical

SUMMARY:
This study investigates whole-body distribution kinetics of intravenously administered Gallium-69 (68Ga) citrate by positron emission tomography (PET)/computed tomography (CT). Thereafter, radiation dosimetry of 68Ga-citrate PET/CT will be determined.

DETAILED DESCRIPTION:
Six healthy male volunteers are recruited in this study. Gallium-68 citrate radiopharmaceutical is intravenously injected as a bolus and whole-body distribution kinetics are studied by dynamic whole-body positron emission tomography/computed tomography. During imaging, serial venous blood samples are drawn, plasma is separated and radioactivity is measured by gamma counter. Immediately after imaging session, urine is voided and radioactivity is measured by gamma counting. As a final point, radiation dosimetry due to single Gallium-68 citrate injection is determined.

ELIGIBILITY:
Inclusion Criteria:

* healthy 18-100 year-old men

Exclusion Criteria:

* ongoing infection/inflammation proven by blood or other tests

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Whole-body distribution of Gallium-68 citrate | 4 hours

SECONDARY OUTCOMES:
Absorbed dose | 4 hours
  Absorbed ionisation radiation dose in critical organs due to intravenous bolus injection of 200 MBq of Gallium citrate

CONTACTS AND LOCATIONS:
Overall Officials: Anne Roivainen, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital/Turku PET Centre, Turku, Finland